CLINICAL TRIAL: NCT06724198
Title: Quality of Life (QoL) and Symptom Burden After Low Rectal Resection. An Open, Effect Pilot Study With Psyllium Husk Treatment in Rectal Cancer Patients.
Brief Title: Bowel Dysfunction After Low Rectal Resection. An Pilot Study Using Psyllium Husk In Rectal Cancer Patients.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Telemark (Other Government)
Responsible Party: Principal Investigator, Silje Stensholt Holte, Principal Ivestigator Consultant Colorectal Surgeon, Sykehuset Telemark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024/732141(REK)
Record Dates: First submitted 2024-11-27; First posted 2024-12-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Low Anterior Resection Syndrome; Quality of Life (QOL)
Keywords: rectal cancer, LARS, quality of life, Psyllium
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms | interventions — Psyllium; Vi-siblin; citric acid, ispaghula husk, sodium bicarbonate drug combination

STUDY DESIGN:
Intervention Model Description: Open-label, effect study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): Participants will recieve Psyllium husk twice daily for 8 weeks
  Interventions: Dietary Supplement: Psyllium husk

INTERVENTIONS:
Dietary Supplement: Psyllium husk — 3.66 gram Psyllium husk twice daily for 8 weeks
  Other Names: Vi-Siblin, Metamucil, Fybogel

SUMMARY:
Rectal cancer constitutes 1/3 of more than 4500 annually diagnosed cases of colorectal (CRC) in Norway. With the advances in radiochemotherapy, and surgical techniques, the long-term survival rate is increasing after surgery regardless of the rising incidences, with a 73% 5-year survival rate in Norway (89% for stage I-III cancer). Low anterior resection (LAR) is the most commonly performed surgical procedure with curative intent with over 500 procedures per year in Norway alone. 80 % of patients subjected to LAR suffer from the LAR syndrome (LARS) which includes grades of bowel incontinence, urgency and tenesmus contributing to reduced quality of life (QoL). Suggested means of management have been advocated without preceding randomized trials. Psyllium husk has been suggested as a nutritional supplement for symptom reduction in patients suffering from LARS, but data is limited and no larger, randomized studies regarding its effect on patients with low anterior resection syndrome have been conducted. In this pilot study preceeding a placebo-controlled RCT, the investigators aim to improve documentation of a proposed management strategy. The investigators anticipate that a reduction in intestinal symptomburden will increase QoL for this large patientgroup.

ELIGIBILITY:
Inclusion Criteria:

* Operated with low rectal resection for rectal cancer
* LARS score >20 at 12 months or more after surgery
* Written consent

Exclusion Criteria:

* Various conditions rendering the patient unable to answer questionnaire
* LARS score 0-20
* Contraindications to Psyllium husk (hypersensitivity, intestinal obstruction, reduced esophageal function, rare congenital medical conditions such as sucrase-isomaltase deficiency, fructose intolerance and glucose-galactose malabsorbtion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
LARS score | At baseline, at 4 and 8 weeks of intervention
  Low anterior resection syndrome score (0-42 points) 0-20: No LARS 21-29: Minor LARS 30-42: Major LARS

SECONDARY OUTCOMES:
Quality of Life (QoL) | At baseline, at 4 and 8 weeks of intervention
  PROMs for self-evaluation of QoL:
  EQ-5D-5L VAS score (0-100 were 0 is the worst possible health and lowest quality of life and 100 is the best possible health and highest quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Silje S Holte, Principal Investigator — Sykehuset Telemark
Locations (1):
- Sykehuset Telemark HF, Skien, Telemark, Norway

IPD SHARING:
Plan to Share IPD: Yes
Results in terms outcomes and patient compliance will be used to stengthen the protocoll for the RCT
Supporting Information: Study Protocol
Time Frame: After study completion
Access Criteria: Collaborators